CLINICAL TRIAL: NCT04740255
Title: Clinical Trial Study for the Use of Straberi Epistamp Needling Device to Treat Postinflammatory Hyperpigmentation (PIH)
Brief Title: Straberi Epistamp Device for Postinflammatory Hyperpigmentation
Acronym: EPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universal Skincare Institute (Other)
Collaborators: Lavish Beauty (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1115
Record Dates: First submitted 2020-09-15; First posted 2021-02-05 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-01

CONDITIONS: Postinflammatory Hyperpigmentation
Keywords: needling; postinflammatory hyperpigmentation; Epistamp; Universal Skincare Institute
MeSH Terms: conditions — Hyperpigmentation | interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Intervention Model Description: Participants in the Straberi by Epistamp device trial, are those who are seeking improvement for Postinflammatory Hyperpigmentation (PIH) caused by acne.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Straberi Epistamp Needling Treatment (Other): Non-Randomized treatment for patients with Postinflammatory Hyperpigmentation (PIH) using the Straberi Epistamp needling.
  Interventions: Device: Straberi Epistamp
- No Treatment (Other): Non-Randomized patients with Postinflammatory Hyperpigmentation (PIH)
  Interventions: Device: Straberi Epistamp

INTERVENTIONS:
Device: Straberi Epistamp — The patient's entire face will be treated. The following settings will be used as a treatment protocol. Needle length between .02- 1.55 mm
  Other Names: Microneedling

SUMMARY:
This pilot study will expand knowledge and application needling using the Straberi device for the improvement of Postinflammatory Hyperpigmentation (PIH) caused by acne.

DETAILED DESCRIPTION:
This pilot study will expand the knowledge and application of needling using the Straberi Epistamp device and its safety and benefits for improving the appearance of Postinflammatory Hyperpigmentation. Postinflammatory Hyperpigmentation (PIH) caused by acne is a common inflammatory disease that can adversely affect facial appearance. Facial acne can have a serious negative impact on psychosocial functioning leaving deep emotional scars. Severe acne can also lead to physical scars and disfigurement. Among patients with severe acne, facial scarring affects both genders equally and occurs to some degree in 95% of cases.

ELIGIBILITY:
Inclusion Criteria:

* Derma Scan showing aging including skin texture, wrinkles, brown spots, and pores.
* Patients willing to sign informed consent.
* Patients willing to be photographed and video documented
* Patients willing to consent to 3 months of treatment

Exclusion Criteria:

* History of eczema in the treatment area; psoriasis and any other chronic skin conditions
* History of actinic (solar) keratosis in the treatment area;
* History of hemophilia
* History of diabetes
* The presence of raised moles, warts on the targeted area.
* Collagen vascular diseases or cardiac abnormalities
* Blood clotting problems
* Active bacterial or fungal infection
* Facial melanosis
* Malignant tumors
* Immunosuppression
* Use of blood thinners or prednisone
* Corticosteroids within two weeks of the procedure
* Chronic liver disease
* Porphyria or other skin diseases.
* Patient not willing to sign informed consent.
* TCA peels in the last 5 weeks
* Subject currently has moderate to severe acne on the face.
* Microneedling within the last 6 months
* Subject has an active infection.
* Subject has a history of a bleeding disorder
* Subject has a history of keloidal tendency
* Subject has received ablative or non-ablative laser treatments in the previous 6 months.
* Subject has taken Accutane within the previous 3 months.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-23 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
The Global Aesthetic Improvement Scale (GAIS) | 6 months
  The Global Aesthetic Improvement Scale (GAIS) is a 5-point scale rating global aesthetic improvement in appearance, compared to pretreatment, as judged by the investigator 5 point scale ranging from 1 to 5 with 5 = The appearance has worsen compared with the original condition and 1 = Excellent corrective results
  compared to pretreatment, as judged by the investigator.

SECONDARY OUTCOMES:
Overall Skin improvement assessed by Derma Scan | 6 months
  The Derma Scan System utilizes two special lighting systems (RGB +UV) and smart skin analyzer software that allows two images (before and after care) to be compared side by side, which can be used to detect the changes in skin
Overall Skin improvement assessed by Post Acne Hyperpigmentation Index (PAHPI) | 6 months
  The parameters of the scoring method are: median lesion size (S) (<3mm, 3-6, 7-10, and >10mm scored as 2, 4, 6, and 8, respectively), median lesion intensity (I) (slightly or moderately or significantly darker than surrounding skin scored as 3, 6, and 9, respectively), and number of lesions (N) (1-15, 16-30, 31-45, 46-60, and >60 scored as 1-5, respectively). The score range from the total of S+I+N=6-22.
Photographs | 6 months
  Digital imaging device using a grid background with controlled lighting and setting to grade acne scar improvement on a quartile grading scale(1 = 1% to 25%, 2 = 26 to 50%, 3 = 51 to 75%, 4 = >76% improvement).
To evaluate the impact on the quality of life (DLQI) | 6 months
  The Dermatology Life Quality Index questionnaire (DLQI) is 10 questions were asked to the patients and score is 0-3 for each question. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.

CONTACTS AND LOCATIONS:
Overall Officials: Maurice E Wright, MD, Principal Investigator — Columbia University; Leslie L Nesbitt, Study Chair — Universal Skincare
Locations (1):
- Lavish, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Once the overall trial is completed and sensitive detailed information is legally advised to published.

REFERENCES:
- [Result] Goodman GJ, Baron JA. Postacne scarring: a qualitative global scarring grading system. Dermatol Surg. 2006 Dec;32(12):1458-66. doi: 10.1111/j.1524-4725.2006.32354.x. PMID 17199653
- [Result] Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol. 1994 May;19(3):210-6. doi: 10.1111/j.1365-2230.1994.tb01167.x. PMID 8033378
- See also: Description Derma Scan — http://universalskincareinstitute.com/
- See also: Description Acne Scars Subtypes — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2958495/